CLINICAL TRIAL: NCT05141084
Title: Weight Loss in Primary Care With Targeted Education and Frequent Follow Ups
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ambereen Ahmed, Integrative Medicine Fellow and Junior Faculty, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aahmed1
Record Dates: First submitted 2021-11-06; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Education, lifestyle — The weight loss program itself is the intervention, which will involve lifestyle modifications and intervention.

SUMMARY:
The investigators will be recruiting patients in the primary care setting to enroll a weight loss program where they will be seen every 2 weeks for 3 months, and then every month for 3 months, and the investigators will implement specific interventions tailored to the patients' needs.

DETAILED DESCRIPTION:
Previous studies have shown that weight loss programs with a multidisciplinary approach in the primary care setting have been more successful in achieving weight loss in overweight and obese patients compared to general recommendations to lose weight. A multidisciplinary approach may include involvement of a dietician and a behavioral psychologist, which the investigators will not be able to replicate in our study. However, some of those studies have also shown that frequent follow-up visits have also been shown to be helpful for weight loss. Frequent follow ups help with weight loss because it helps patients maintain their accountability by giving them realistic goals with measurable deadlines. Education is also an important factor to weight loss, including understanding an individualized dietary and exercise approach. Weight loss in the primary care setting is of great significance because it can offload healthcare costs by reducing the morbidity of disease for a variety of comorbid conditions such as diabetes, hypertension or hyperlipidemia. Studies have shown that exercise alone (without any reduction in weight) improves hypertension and glucose sensitivity in patients. The investigators hypothesize that achieving weight loss will have an additive effect to these health improvements. The American Heart Association recently revised their cholesterol guidelines for reducing atherosclerotic cardiovascular disease (ASCVD) by listing the first and foremost recommendation as: "a healthy lifestyle reduces ASCVD risk at all ages. In all age groups, lifestyle therapy is the primary intervention for metabolic syndrome." So, diet and lifestyle modifications are recognized by many societies as an important and necessary intervention for patients to live healthy lives and decrease the morbidity and mortality associated with disease.

Additionally, overweight and obese people also have a high incidence of chronic joint pains which often result in therapies, invasive joint surgeries, immobility, or chronic treatments with prescription pain medications. It has been shown that these joint pains can be reduced with weight loss preventing the need for those aforementioned therapies which have a high cost burden on the healthcare system. The biggest determining factor of weight loss is a person's adherence to the intervention, which will hope to address with close follow up to hold patient's accountable to their weight loss goals.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30
* English and Spanish speaking
* All ethnicities

Exclusion Criteria:

* Those who have had bariatric surgery within the last 1 year or are actively still losing weight from bariatric surgery
* Those who are part of another weight loss program
* Those who are actively using substances such as drugs or alcohol
* Pregnant women
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Weight | through study completion, anticipated 6 months
Waist circumference | through study completion, anticipated 6 months
Body fat percentage | through study completion, anticipated 6 months

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | through study completion, anticipated 6 months
Hemoglobin a1c | through study completion, anticipated 6 months
Cholesterol | through study completion, anticipated 6 months
Patient Health Questionnaire-9 | through study completion, anticipated 6 months
  Measure of depression, maximum score of 27 indicating severe depression, minimum score of 0 indicating likely no depression
Generalized Anxiety Disorder-7 | through study completion, anticipated 6 months
  Measure of anxiety, maximum score of 21 indicating severe anxiety, minimum score of 0 meaning likely no anxiety

IPD SHARING:
Plan to Share IPD: No